CLINICAL TRIAL: NCT05463848
Title: A Surgical "Window-of-Opportunity" and Phase II Trial of Pembrolizumab, Olaparib and Temozolomide in Recurrent Glioblastoma
Brief Title: Surgical Pembro +/- Olaparib w TMZ for rGBM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: L. Nicolas Gonzalez Castro, MD, PhD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, L. Nicolas Gonzalez Castro, MD, PhD, Sponsor-Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-251; MISP 60154 (Other: Merck & Co., Inc.)
Record Dates: First submitted 2022-07-12; First posted 2022-07-19 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma; Recurrent Glioblastoma
Keywords: Glioblastoma; Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — pembrolizumab; olaparib; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Safety Lead In): pembrolizumab plus olaparib and temozolomide (Experimental): Following a 3 + 3 dose escalation design 6-18 participants will receive:
  * Olaparib 2x daily on Days 1-7 of each 21-day study cycle.
  * Temozolomide 1x daily on Days 1-7 of each 21-day study cycle.
  * Pembrolizumab on Day 1 of every other 21-day cycle (once every 6 weeks).
  Interventions: Drug: Pembrolizumab; Drug: Olaparib; Drug: Temozolomide
- Cohort 2 (Surgical Cohort): Arm A - Pembrolizumab plus olaparib and temozolomide (Experimental): Cohort 2 participants will be randomized into either group a or b (1:1):
  Group A participants will receive pembrolizumab, olaparib, and temozolomide before and after surgery.
  * Olaparib 2x daily on Days 1-7 of each 21-day study cycle.
  * Temozolomide 1x daily on Days 1-7 of each 21-day study cycle.
  * Pembrolizumab on Day 1 of every other 21-day cycle (once every 6 weeks).
  Interventions: Drug: Pembrolizumab; Drug: Olaparib; Drug: Temozolomide
- Cohort 2 (Surgical Cohort): Arm B - Pembrolizumab monotherapy (Experimental): Cohort 2 participants will be randomized into either group a or b (1:1):
  Group B participants will receive pembrolizumab monotherapy before and after surgery.
  * Pembrolizumab Before Surgery: Day 1 of the pre-surgical treatment cycle.
  * Pembrolizumab After Surgery: Day 1 of every other 21-day cycle (once every 6 weeks).
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Intravenous infusion
  Other Names: MK3475
Drug: Olaparib — Pill taken by mouth
  Other Names: MK-7339
  Arms: Cohort 1 (Safety Lead In): pembrolizumab plus olaparib and temozolomide; Cohort 2 (Surgical Cohort): Arm A - Pembrolizumab plus olaparib and temozolomide
Drug: Temozolomide — Pill taken by mouth
  Other Names: Temodar
  Arms: Cohort 1 (Safety Lead In): pembrolizumab plus olaparib and temozolomide; Cohort 2 (Surgical Cohort): Arm A - Pembrolizumab plus olaparib and temozolomide

SUMMARY:
This research study is studying a combination therapy as a possible treatment for recurrent glioblastoma (GBM), a brain tumor that is growing or progressing despite earlier treatment.

The names of the study interventions involved in this study are/is:

* Pembrolizumab
* Olaparib
* Temozolomide (Temodar)

DETAILED DESCRIPTION:
This is an open label, multi-center, phase II trial evaluating the safety and efficacy of olaparib, temozolomide and pembrolizumab in participants with recurrent glioblastoma at their first or second relapse.

The U.S. Food and Drug Administration (FDA) has not approved pembrolizumab or olaparib for recurrent glioblastoma, but both have been approved for other uses.

Pembrolizumab is an antibody designed to block the action of the receptor, PD-1. PD-1 works to help tumor cells inhibit the immune system's response against a tumor. Olaparib is an inhibitor of PARP (poly [adenosine diphosphate-ribose] polymerase) an enzyme found in the cells of the human body that helps cells, including cancer cells, survive and grow by repairing DNA damage in the cells. Olaparib helps kill cancer cells by preventing PARP from repairing their DNA.

The U.S. FDA has approved temozolomide as a treatment option for glioblastoma. Temozolomide is a chemotherapy drug that can enter the brain and prevent tumor cells from growing by causing DNA damage.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

It is expected that all participants will receive pembrolizumab for up to 2 years or as long as they do not have serious side effects and their disease does not get worse. It is expected that Cohort 1 and Cohort 2 Arm A participants will receive Olaparib and temozolomide for as long as they do not have serious side effects and their disease does not get worse.

It is expected that about 66-78 people will take part in this research study.

Merck Sharp & Dohme Corp., a subsidiary of Merck & Co., Inc., is supporting this research study by providing funding for the research study and both investigational study drugs, pembrolizumab and olaparib.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to understand and willing to sign a written informed consent document.
* Participants must be able to adhere to the dosing and visit schedules and agree to record medication times accurately and consistently in a daily diary.
* Participants must be at least 18 years old on day of signing informed consent.
* Women of childbearing potential are eligible to participate if they are not pregnant or breastfeeding.
* Participants must have a Karnofsky Performance Status (KPS) ≥ 70 and Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1 (see Appendix A).
* Participants must be able to swallow oral medications. Nature of illness and treatment history
* Participants must have histologically World Health Organization Grade IV IDH wildtype glioblastoma by IDHR132H immunohistochemistry or variants including gliosarcoma or IDH wildtype diffuse glioma with molecularly features of glioblastoma (EGFR amplification, TERT promoter mutation, or concurrent gain of Chromosome 7 and loss of Chromosome 10) (Brat et al., 2018). IDH mutational status can be established via immunohistochemistry and/or next-generation sequencing.
* Participants must be at first or second relapse of GBM. First relapse is defined as progression following initial therapy and second relapse is progression following second therapy. The intent therefore is that patients had no more than 2 prior therapies (i.e. radiation +/- chemotherapy if that was used as initial therapy and one additional therapy for first recurrence). If the patient had a surgical resection for relapsed disease and no anti-cancer therapy was instituted for up to 12 weeks, and the patient undergoes another surgical resection, this is considered to constitute 1 relapse.
* Participants must have shown unequivocal evidence for tumor progression by MRI scan per modified RANO criteria (Ellingson et al., 2017).
* MRI should be obtained within 14 days prior to study registration.
* Confirmation of availability of sufficient tissue from a prior surgery demonstrating glioblastoma for correlative studies is required prior to enrollment.

  * Cohort 1: 15 unstained FFPE sections (standard 10 micrometer thickness)
  * Cohort 2: 1 (FFPE) block (preferred) OR 35 unstained FFPE sections (standard 5 micrometer thickness)
  * NOTES:

    * If the above-mentioned tissue is not available from the most recent surgery revealing GBM, participants may be enrolled with tissue available from any prior surgery revealing GBM with prospective approval from the Principal Investigator.
    * If the participant's slides have been reviewed on a previous study and there has been no interim surgery or biopsy, slides do not need to be re-submitted for histologic confirmation. The site must submit a copy of the previous submission forms with the review results to the central office as documentation for the new study.
* Cohort 2 patients only: Surgically resectable disease at progression.

  * There must be > 2cm3 enhancing tissue available for resection and submission for study correlatives as determined by local treating team.
  * For the first 10 patients in Arm A who will have tumor resected for analysis of olaparib levels, both enhancing and non-enhancing tumor should be available for resection.
* An interval of at least 12 weeks from the completion of radiation therapy to start of study drug unless there is unequivocal histologic confirmation of tumor progression.
* Participants must have recovered to grade 0 or 1 or pre-treatment baseline from clinically significant toxic effects of prior therapy (including but not limited to exceptions of alopecia, laboratory values listed per inclusion criteria, and lymphopenia which is common after therapy with temozolomide).
* An interval of at least 4 weeks (to registration) between prior surgical resection or one week for stereotactic biopsy.
* From registration the following time periods must have elapsed (some previous therapies are exclusionary; see items 26-29 under Exclusion Criteria):

  * 4 weeks or 5 half-lives (whichever is shorter) from any investigational agent;
  * 4 weeks from cytotoxic therapy (except 23 days for temozolomide; 6 weeks from nitrosoureas);
  * 4 weeks or 5 half-lives (whichever is shorter) from antibodies;
  * 4 weeks or 5 half-lives (whichever is shorter) from other anti-tumor therapies.
  * No washout required for tumor treating fields.

Clinical labs - Participants should have adequate organ function, in accordance to the studies outlined below. All screening laboratory tests should be performed within 10 days prior to the first dose of the study intervention.

* Hematology:

  * Leukocytes ≥ 3,000/µL
  * Absolute neutrophil count (ANC) ≥ 1,500/µL
  * Platelet count ≥ 100,000/µL
  * Absolute Lymphocyte Count ≥ 500/µL
  * Hemoglobin ≥ 9.0 g/dL
* Biochemistry:

  * AST (SGOT) and ALT (SGPT) ≤ 2.5 x institution's ULN (or ≤ 5 X institutional ULN for subjects with Gilberts syndrome)
  * Serum bilirubin ≤ 1.5 x institution's ULN or direct bilirubin ≤ institutional ULN for subjects with total bilirubin levels > 1.5 institutional ULN.
  * Serum creatinine ≤ 1.5 x institution's ULN or calculated 24-hour creatinine clearance > 50 mL/min
  * Serum albumin ≥ 2.5 g/dL
  * Coagulation studies:
  * INR ≤ 1.5 X institutional ULN
  * PTT ≤ institution's ULN, unless receiving therapeutic low molecular weight heparin or oral factor Xa inhibitors.

Other illnesses

* History of known additional malignancy that is progressing or requires active treatment. Those patients whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen will be eligible including, but not limited to, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, localized prostate cancer not requiring treatment, or in situ cervical cancer that has undergone potentially curative therapy.

Pregnancy and Reproduction

* Olaparib has been shows to be teratogenic in rats. The effects of pembrolizumab on the developing human fetus are unknown. For this reason:

  * Female Participants:

    * A female patient is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies:

      * Not a woman of childbearing potential (WOCBP) as defined in Appendix L OR
      * A WOCBP who agrees to follow the contraceptive guidance in Appendix L during the treatment period and for at least 120 days after the last dose of study intervention, corresponding to time needed to eliminate any study intervention(s) (ie, olaparib) plus 30 days (a menstruation cycle) for study interventions with risk of genotoxicity.
    * Women of child-bearing potential (WOCBP) must have a negative serum or urine β human chorionic gonadotropin (β-hCG) pregnancy test within 7 days prior to first dose of olaparib and/or pembrolizumab. (NOTE: Pregnancy test will be repeated within 72 hours prior to Day 1 drug if original screening pregnancy test is not within 72 hours of Day 1 drug.)
  * Male Participants: A male patient must agree to use contraception as detailed in Appendix L of this protocol during the treatment period and for at least 180 days, corresponding to time needed to eliminate any study intervention(s) (ie, olaparib) plus a spermatogenesis cycle, after the last dose of study intervention and refrain from donating sperm during this period.

Exclusion Criteria:

Pathology

* Prior evidence of 1p/19q co-deletion.
* IDH mutation by immunohistochemistry or by sequencing.
* Tumor primarily localized to the brainstem or spinal cord.
* Presence of diffuse leptomeningeal disease or extracranial disease.

Previous therapies

* Participants who have received prior treatment with a PARP inhibitor (e.g. olaparib, niraparib).
* Participants who have received anti-VEGF targeted agents (e.g. bevacizumab, cediranib, aflibercept, vandetanib, cabozantinib, sunitinib etc.).
* Participants who have received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Participants who have received prior viral therapy or vaccines for glioblastoma.
* Participant received colony-stimulating factors (e.g., granulocyte colony-stimulating factor [G-CSF0], granulocyte-macrophage colony-stimulating factor [GM-CSF] or recombinant erythropoietin) within 28 days prior to the first dose of study intervention.

Concomitant medications

* Participants requiring treatment with high dose systemic corticosteroids defined as dexamethasone > 2 mg/day or bioequivalent for at least 3 consecutive days within 2 weeks of start of study drug.
* Participants who have received systemic immunosuppressive treatments, aside from systemic corticosteroids (such as methotrexate, chloroquine, azathioprine, etc.) within six months of start of study drug.
* Participants taking an enzyme-inducing anti-epileptic drug (EIAED): phenobarbital, phenytoin, fosphenytoin, primidone, carbamazepine, oxcarbazepine, eslicarbazepine, rufinamide, and felbamate. Participants must be off any EIAEDs for at least 14 days prior to starting study drug. A list of EIAEDs and other inducers of CYP3A4 can be found in Appendix D. Among non-EIAED, caution is recommended with use of valproic acid due to potential for drug interaction.
* Participants taking a drug known to be a strong inhibitor or inducer of isoenzyme CYP3A (Appendix D). Participant must be off CYP3A inhibitors and inducers for at least 7 days prior to starting study drug. NOTE: participants must avoid consumption of Seville oranges (and juice), grapefruits or grapefruit juice, grapefruit hybrids, pummelos and exotic citrus fruits from 7 days prior to the first dose of study drug and during the entire study treatment period due to potential CYP3A4 interaction.
* Participants receiving any other investigational agents.
* Current use of herbal preparations/medications, including but not limited to: Cannabinoids, St. John's wort (tablet or tea), Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, ginseng. Participants should stop using these herbal medications 7 days prior to first dose of study drug.
* Current use of warfarin sodium or any other coumadin-derivative anticoagulant. Participants must be off Coumadin-derivative anticoagulants for at least 7 days prior to starting study drug. Low molecular weight heparin and Factor Xa inhibitors are allowed.

Other illnesses

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to olaparib, temozolomide and/or pembrolizumab.
* History of myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or with features suggestive of MDS/AML.
* History of intratumoral or peritumoral hemorrhage if deemed significant by the treating investigator. If there are questions, the treating investigator should contact the study Principal Investigator, Patrick Y Wen, MD, at 617-632-2166.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, chronic liver disease (e.g., cirrhosis, hepatitis), chronic renal disease, pancreatitis, chronic pulmonary disease, or psychiatric illness/social situations that would limit compliance with study requirements. Subjects must be free of any clinically relevant disease (other than glioma) that would, in the treating investigator's opinion, interfere with the conduct of the study or study evaluations.
* Participant has an active infection requiring systemic therapy and/or known viral infection (for example, human immunodeficiency virus antibodies, hepatitis B surface antigen or hepatitis C antibodies).
* Participant with a known history of active TB (Bacillus Tuberculosis).
* Participant with a diagnosis of immunodeficiency, including a known history of Human Immunodeficiency Virus (HIV).
* Participant with active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Participants who have received a live vaccine within 30 days prior to start of study treatment. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, BCG, and typhoid vaccine.

Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

* Participants with diarrhea ≥ CTCAE grade 2
* Participant has active cardiac disease including any of the following:

  * Angina pectoris that requires the use of anti-anginal medications.
  * Ventricular arrhythmias except for benign premature ventricular contractions.
  * Supraventricular and nodal arrythmias requiring a pacemaker or not controlled with medication.
  * Conduction abnormality requiring a pacemaker.
  * Valvular disease with document compromise in cardiac function.
  * Symptomatic pericarditis.
  * Unstable ischemia
  * QTc prolongation >500 ms (calculated via the Fridericia formula)
  * Electrolyte disturbances
* Participant has a history of cardiac dysfunction including any of the following:

  * Myocardial infarction within the last 6 months prior to start of study drug, documents by persistent elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LVEF function.
  * History of documented congestive heart failure (New York Heart Association functional classification III-IV, see Appendix K).
  * Documented cardiomyopathy.
  * Congenital long QT syndrome.
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of olaparib and temozolomide (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or extensive small bowel resection). Participants with unresolved diarrhea ≥ CTCAE grade 2 will be excluded as previously indicated.
* Participants who have undergone major systemic surgery < 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
* Participants who are pregnant or breastfeeding.
* Participants with history of known coagulopathy that increases risk of bleeding or a history of clinically significant hemorrhage within 12 months of start of study drug or gastrointestinal bleeding or any other hemorrhage/bleeding event CTCAE Grade > 3 within 6 months of start of study drug.
* Has known history of, or any evidence of, active non-infectious pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-10-21 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Tumor infiltrating lymphocytes (TIL) Density | At surgery. Surgery will occur 14 days +/- 5 days after initiation of treatment.
  TIL density quantifies anti-tumor immune response. It is measured in tumor tissue from protocol surgery, analyzed by immunohistochemistry and by next generation sequencing.
6-month Progression-Free Survival (PFS6) | 6 months after surgery. Surgery will occur 14 days +/- 5 days after initiation of treatment.
  Progression-free survival based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) or death. PD defined by modified RANO as well as iRANO criteria, per protocol section 12.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 24 months
  The objective response rate (ORR) was defined as the proportion of participants achieving complete response (CR) or partial response (PR) based on modified RANO as well as iRANO criteria, per protocol section 12.
Median Overall Survival (OS) | 24 months
  OS based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.
Grade 3 or Higher Treatment-Related Toxicity Rate | 24 months
  All grade 3 or higher adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv5 as reported on case report forms were counted. Rate is the proportion of treated participants experiencing at least one treatment-related grade 3 or higher AE of any type during the time of observation.
Gene expression profiling (GEP) score | At surgery. Surgery will occur 14 days +/- 5 days after initiation of treatment.
  GEP score uses surgery tumor tissue to measure cell-cycle related gene signatures in the tumor microenvironment per established methods.

CONTACTS AND LOCATIONS:
Overall Officials: Luis N Gonzalez Castro, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu